CLINICAL TRIAL: NCT07286357
Title: A Multi-Center Retrospective Data Collection Protocol to Evaluate the Real World Usage of the Orthofix AccelStim Device to Treat Fresh Metatarsal Fractures
Brief Title: A Data Collection Protocol to Evaluate the Real World Usage of the Orthofix AccelStim Device to Treat Fresh Metatarsal Fractures
Acronym: ASRW
Status: Active, not recruiting | Type: Observational
Sponsor: Orthofix Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP-ASRW-24
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Metatarsal Fracture

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- AccelStim (LIPUS): This group will include subjects where AccelStimStim (LIPUS) is used to treat fresh metatarsal fracture
  Interventions: Device: AccelStim (LIPUS)
- Control (no LIPUS device): This group will include subjects where AccelStimStim (LIPUS) was not used to treat fresh metatarsal fracture

INTERVENTIONS:
Device: AccelStim (LIPUS) — Subjects treated with LIPUS were directed to use the AccelStim device for 20 minutes per day, up to 6 months or until no longer needed.
  Other Names: Low Intensity Pulsed UltraSound
  Groups: AccelStim (LIPUS)

SUMMARY:
This study examines the effect of using the AccelStim bone growth stimulator on subjects undergoing treatment for fresh metatarsal fractures.

DETAILED DESCRIPTION:
The objective of this investigation is to study the effect of using LIPUS treatment (via AccelStim) in subjects with fresh metatarsal fractures. The sponsor hypothesizes that use of AccelStim will result in higher rates of fusion compared to that of control. In addition to analyzing the primary endpoint, the study will collect safety information to confirm the favorable safety profile established in prior device usage.

ELIGIBILITY:
Inclusion Criteria:

* Fresh metatarsal fracture patient that has been prescribed an Orthofix AccelStim device
* Patient is 18 years or older at the time of treatment

Exclusion Criteria:

-Patient is a prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who were treated for eligible fresh metatarsal fractures and were subsequently prescribed an Orthofix AccelStim device will be considered for participation in this retrospective study. Cases will be identified by searching local medical records and/or device prescription information received at Orthofix.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Healing Status | 3, 6, and 12 month
  Quantitative and qualitative assessments of clinical and radiographic healing (as available per standard of care)

SECONDARY OUTCOMES:
Pain (NPRS) (0-100) | Baseline, 3, 6, and 12 month
  Numerical Pain Rating Scale (NPRS) (0-100, where 100 is maximum pain)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Northwestern, Evanston, Illinois
  - Endeavor Health, Mount Prospect, Illinois
  - Precision Orthopedics, Laurel, Maryland

IPD SHARING:
Plan to Share IPD: No